CLINICAL TRIAL: NCT04272203
Title: A Phase 1 First in Human, Multicenter, Open-Label Dose-Escalation Study to Determine the Safety, Tolerability, Pharmacokinetics, and RP2D of ABBV-184 in Subjects With Previously Treated Cancers
Brief Title: A Study to Determine Safety, Tolerability, Pharmacokinetics, and Recommended Phase 2 Dose (RP2D) of Intravenous ABBV-184 in Adult Participants With Previously Treated Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M19-747; 2019-003434-16 (EudraCT Number)
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia (AML); Non Small Cell Lung Cancer; Cancer
Keywords: Advanced Solid Tumors Cancer; Acute Myeloid Leukemia (AML); Non Small Cell Lung Cancer (NSCLC); Blood Cancer; ABBV-184; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Carcinoma, Non-Small-Cell Lung; Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose Escalation: Participants With AML (Experimental): Participants with relapsed or refractory (R/R) AML will receive escalating doses of ABBV-184
  Interventions: Drug: ABBV-184
- Dose Escalation: Participants With NSCLC (Experimental): Participants with relapsed or refractory (R/R) NSCLC will receive escalating doses of ABBV-184
  Interventions: Drug: ABBV-184
- Dose Expansion: Participants With AML (Experimental): Participants with R/R AML will receive ABBV-184 at recommended Phase 2 dose (RP2D) determined in dose escalation phase for AML
  Interventions: Drug: ABBV-184
- Dose Expansion: Participants With NSCLC (Experimental): Participants with R/R NSCLC will receive ABBV-184 at RP2D determined in dose escalation phase for NSCLC
  Interventions: Drug: ABBV-184

INTERVENTIONS:
Drug: ABBV-184 — Intravenous (IV) infusion

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. This study focuses on two types of cancers: Acute Myeloid Leukemia (AML) and Non-Small Cell Lung Cancer (NSCLC). AML (blood cancer) is cancer of the white blood cells (WBC). NSCLC (solid tumor) is a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to determine recommended phase 2 dose (RP2D) and to see if the study drug is safe and able to treat patients who have AML and NSCLC.

ABBV-184 is an investigational drug being developed for treatment of cancer. The study has two arms and two phases: AML arm and NSCLC arm; dose escalation and dose expansion phase. Adult participants with diagnosis of AML or NSCLC will be enrolled. In dose escalation phase, around 36 participants will be enrolled in each arm. In dose expansion phase, around 20 participants will be enrolled in each arm. The study will be conducted in approximately 50 sites across 10 countries.

Participants will receive weight based intravenous (IV) infusion of ABBV-184 once a week. At the beginning of the study, visits will occur daily during hospitalization followed by less frequently over time.

There will be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of treatment will be checked by medical assessments, blood tests, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) or non-small cell lung cancer (NSCLC).
* Participants must consent to hospitalization for at least 72 hours following the first two doses of ABBV-184 in Cycle 1.
* Participants must have Human Leukocyte Antigen-A2 (HLA-A2) restricted genotype. Participants must be HLA-A2:01 positive in at least one allele tested with a high-resolution HLA genotyping assay performed in a College of American Pathologists (CAP)/Clinical Laboratory Improvement Act (CLIA)-certified or equivalent laboratory.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Laboratory values and cardiac function must meet the protocol specifications.

Exclusion Criteria:

* For AML participants:

  * Presence or history of extramedullary disease are ineligible, participants with a diagnosis of acute promyelocytic leukemia (APL) or BCR-ABL-positive leukemia are not eligible.
* For NSCLC participants:

  * Tumors with epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) gene rearrangements are not eligible.
* Active/uncontrolled central nervous system (CNS) leukemia/lung cancer are not eligible for the study.
* History of inflammatory bowel disease, interstitial lung disease (pneumonitis), myocarditis, Stevens-Johnson syndrome, toxic epidermal necrolysis, solid organ transplantation, active autoimmune disease (with exceptions of vitiligo, Type I diabetes mellitus, hypothyroidism, and psoriasis), primary immunodeficiency.
* History of clinical diagnosis of tuberculosis or major immunologic reaction to any immunoglobulin G (IgG)-containing agent are not eligible.
* Previously received anti-cancer treatment with an agent that targets the immune system by engaging cluster of differentiation 3 (CD3) are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of ABBV-184 (Dose-Escalation Phase) | Up to 1 Cycle after the last participant is enrolled in dose escalation phase (Approximately 2 years)
  The RP2D of ABBV-184 will be determined during the dose-escalation phase of the study. RP2D will be determined using available safety and pharmacokinetics and pharmacodynamics data.
Complete Remission (CR) or Complete Remission With Partial Hematologic Recovery (CRh) Rate (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  CR/CRh rate is assessed based on the Clopper-Pearson (exact) method.
Objective Response Rate (ORR) (Dose Expansion Phase in Participants With NSCLC) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  ORR is defined as participants with confirmed complete or partial response (CR+PR) per RECIST, v1.1

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Change in Laboratory Parameters | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Number of participants with clinically significant change from baseline in clinical laboratory test results like hematology will be reported.
Change in Vital Signs | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Number of participants with clinically significant change from baseline in vital signs like systolic and diastolic blood pressure will be reported.
Change in Montreal Cognitive Assessment (MoCA) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  The Montreal Cognitive Assessment (MoCA) is a one page 30-point written test that assesses cognitive function.
Change in Echocardiogram | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Number of participants with abnormal change from baseline in echocardiogram will be reported.
Change in Electrocardiogram (ECG) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  12-lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.
Maximum Observed Serum Concentration (Cmax) of ABBV-184 | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Maximum Serum Concentration (Cmax) of ABBV-184.
Time to Maximum Observed Serum Concentration (Tmax) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Time to Maximum Serum Concentration (Tmax) of ABBV-184.
Terminal Phase Elimination Rate Constant (β) for ABBV-184 | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Terminal Phase Elimination Rate Constant (β) for ABBV-184.
Terminal Phase Elimination Half-life (t1/2) of ABBV-184 | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Terminal Phase Elimination Half-life (t1/2) of ABBV-184.
Area Under the Serum Concentration-Time Curve of ABBV-184 | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Area Under the Serum Concentration-Time Curve of ABBV-184.
Percentage of Participants With Anti-drug Antibodies (ADAs) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Percentage of Participants With Anti-drug Antibodies (ADAs)
Duration of Response (DOR) (Dose Expansion Phase) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  DOR is defined as the time between date of first response and the first occurrence of progression or death from any cause, whichever occurs first.
Progression-free Survival (PFS) (Dose Expansion Phase) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  PFS will be defined as the time between the first dose of any study drug and the first occurrence of progression or death from any cause.
Relapse-Free Survival (RFS) (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  RFS is defined as the time between date of first response and the first occurrence of progression or death from any cause, whichever occurs first.
Change in Bone Marrow Blast Count (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Percentage of blast cells in bone marrow.
Change in Peripheral Blood Blast Count (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  Percentage of blast cells in peripheral blood.
Objective Response Rate (ORR) (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  ORR is defined as the proportion of participants with complete remission (CR), morphologic complete remission with incomplete blood count recovery (CRi), complete remission with partial hematologic recovery (CRh), complete response with incomplete platelet recovery (CRp), and partial remission (PR).
Rate of Conversion to Transfusion Independence (Dose Expansion Phase in Participants With AML) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  AML participants will be considered to have converted to transfusion independence if they receive no red blood cell transfusion, platelet transfusion, or growth factors for a 56-day window after beginning study treatment.
Clinical Benefit Rate (CBR) (Dose Expansion Phase in Participants With NSCLC) | Up to 30 days after last participant complete study drug (Approximately 3 years)
  CBR is defined as the proportion of participants with a CR, PR, or stable disease (SD) for at least 6 weeks by RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (17):
- United States (3):
  - Fort Wayne Medical Oncology and Hematology, Inc /ID# 224332, Fort Wayne, Indiana
  - Gabrail Cancer Center Research /ID# 215667, Canton, Ohio
  - Thomas Jefferson University /ID# 218403, Philadelphia, Pennsylvania
- France (5):
  - Centre Antoine Lacassagne - Nice /ID# 218014, Nice, Alpes-Maritimes
  - CHU Bordeaux - Hopital Haut Leveque /ID# 224998, Pessac, Gironde
  - CHRU Lille - Hopital Claude Huriez /ID# 217508, Lille, Hauts-de-France
  - CHU de Nantes, Hotel Dieu -HME /ID# 215703, Nantes, Pays de la Loire Region
  - Hopital Saint-Andre /ID# 224218, Bordeaux
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 215810, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 222749, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 215808, Haifa
- Japan (3):
  - Aichi Cancer Center Hospital /ID# 216469, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 216467, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 216466, Chuo-ku, Tokyo
- United Kingdom (3):
  - Oxford University Hospitals NHS Foundation Trust /ID# 217252, Oxford, Oxfordshire
  - Cardiff & Vale University Health Board /ID# 217250, Cardiff, Wales
  - The Christie Hospital /ID# 216118, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterlin P, Saada-Bouzid E, Moskovitz M, Pigneux A, Yuda J, Sinnollareddy M, Henner WR, Chen D, Freise KJ, Leibman RS, Avigdor A, Shimizu T. First-in-human clinical trial results with ABBV-184, a first-in-class T-cell receptor/anti-CD3 bispecific protein, in adults with previously treated AML or NSCLC. Expert Rev Anticancer Ther. 2024 Sep;24(9):893-904. doi: 10.1080/14737140.2024.2373888. Epub 2024 Jul 10. PMID 38946484